CLINICAL TRIAL: NCT01222884
Title: A Phase III, Randomized, Comparative, Open-label Study of Intravenous Iron Isomaltoside 1000 (Monofer®) Administered as Maintenance Therapy by Single or Repeated Bolus Injections in Comparison With Intravenous Iron Sucrose in Subjects With Stage 5 Chronic Kidney Disease on Dialysis Therapy (CKD-5D)
Brief Title: A Randomized, Comparative, Open-label Study of IV Monofer® Administered as Maintenance Therapy by Single or Repeated Bolus Injections in Comparison With IV Iron Sucrose in Subjects With CKD-5D
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmacosmos A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-Monofer-CKD-03
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Results first posted 2015-07-24 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Kidney Disease Stage 5 (Dialysis Dependent)
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Ferric Oxide, Saccharated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iron isomaltoside 1000 (Active Comparator): Iron isomaltoside 1000 (Monofer)administered as 500 mg intravenous single bolus injections OR administered as 500 mg fractionated (100mg+200mg+200mg) intravenous bolus injection
  Interventions: Drug: Monofer
- Iron sucrose (Active Comparator): Iron sucrose administered as 500 mg fractionated (100mg+200mg+200mg) intravenous bolus injection
  Interventions: Drug: Iron sucrose

INTERVENTIONS:
Drug: Monofer — Iron isomaltoside 1000 (Monofer®) administered as 500 mg intravenous single bolus injection over approximately 2 minutes
  Arms: Iron isomaltoside 1000
Drug: Iron sucrose — Iron sucrose is administered undiluted in doses of 100mg at baseline, 200mg at week 2 and 200 mg at week 4 as fractionated IV bolus injections according to local Summary of Product Characteristics
  Arms: Iron sucrose

SUMMARY:
The purpose of this study is to compare the efficacy and safety of intravenous iron isomaltoside 1000 with intravenous iron sucrose in patients suffering from Stage 5 Chronic Kidney Disease on Dialysis Therapy (CKD-5D).

ELIGIBILITY:
Inclusion Criteria:

Subjects with a diagnosis of CKD-5D, in dialysis therapy for at least 90 days prior to inclusion, will be included if they meet all of the following criteria:

1. Men or women, aged 18 years or greater.
2. Subjects diagnosed with CKD-5D and in haemodialysis therapy for at least 90 days.
3. Life expectancy beyond 12 months by Principal Investigator's judgement.
4. Willingness and ability to participate after Informed Consent.
5. Hb concentrations between 9.5 g/dL and 12.5 g/dL (both values included) both at Screening Visit 1a and at Screening Visit 1b (screening Visit 1a and Visit 1b must be separated by at least 1 week).
6. Serum ferritin < 800 ng/mL.
7. Transferrin Saturation < 35%.
8. Subjects receiving ESA treatment with dose stable for the previous 4 weeks prior to screening (with only 1 missed dose to be allowed. Dose to be kept stable during the study period).
9. Subjects receiving no IV iron or an average of no more than 100 mg/week for the previous 4 weeks (with only 1 missed dose to be allowed).

Exclusion Criteria:

1. Anaemia caused primarily by factors other than renal related anaemia.
2. Iron overload or disturbances in utilization of iron (e.g. haemochromatosis and haemosiderosis).
3. Patients currently undergoing treatment with immunosuppresives (low dose steroids are allowed during the study conduct for dosages no more than 10 mg prednisolone/day or equivalent. If possible the dosage should be kept constant through the study).
4. Difference of Hb ≥ 1.0 g/dL between screening (Visits 1a and 1b).
5. Patients with a history of multiple allergies.
6. Decompensated liver cirrhosis or active hepatitis [Alanine Aminotransferase (ALT) > 3 times normal] or history of Hepatitis B or C.
7. Active acute or chronic infections (assessed by clinical judgement), supplied with White Blood Cells (WBC) and C - reactive protein (CRP).
8. Rheumatoid arthritis with symptoms or signs of active joint inflammation.
9. Pregnancy or nursing. [To avoid pregnancy, women have to be postmenopausal (at least 12 months must have elapsed since last menstruation), surgically sterile, or women of child bearing potential must use one of the following contraceptives during the whole study period and after the study has ended for at least 5 times plasma biological half-life of the investigational medicinal product: Contraceptive pills, Intrauterine Devices (IUD), contraceptive depot injections (prolonged-release gestagen), subdermal implantation, vaginal ring, and transdermal patches]
10. Blood transfusion within the previous 12 weeks.
11. Planned elective surgery in the next 8 weeks.
12. Participation in any other clinical trial within the past 30 days, or if longer, where the study drug has not passed five half-lives prior to screening.
13. Untreated Vitamin B12 or folate deficiency.
14. Any other medical condition that, in the opinion of Principal Investigator, may cause the subject to be unsuitable for the completion of the study or place the subject at potential risk from being in the study. Examples include Uncontrolled Hypertension, Unstable Ischemic Heart Disease or Uncontrolled Diabetes Mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2011-06; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Lykke Thomsen, MD, Study Chair — Pharmacosmos A/S
Locations (1):
- Jatin Kothari, Mumbai, India

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Iron Isomaltoside 1000 | Iron Sucrose
Started | 234 | 117
Completed | 210 | 113
Not Completed | 24 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Iron Isomaltoside 1000 | Iron Sucrose | Total
Number analyzed (Participants) | 234 | 117 | 351
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 129 | 66 | 195
  >=65 years | 105 | 51 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (16.2) | 59.5 (15.4) | 60.0 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 43 | 119
  Male | 158 | 74 | 232
Region of Enrollment [Number; unit: participants]
  India | 44 | 28 | 72
  United Kingdom | 131 | 56 | 187
  Russian Federation | 6 | 3 | 9
  Poland | 10 | 3 | 13
  Sweden | 6 | 4 | 10
  Switzerland | 13 | 6 | 19
  Romania | 14 | 12 | 26
  Denmark | 6 | 5 | 11
  United States | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Ability to Maintain Hemoglobin Level
Description: The primary outcome measure was the proportion of subjects who were able to maintain haemoglobin between 9.5 and 12.5 g/dL (both values included) at week 6. Haemoglobin was measured by a blood sample at the different visits. All blood samples were taken before the dialysis from the dialysis catheter. Intravenous iron was administered during dialysis, at least 30 min after the start and at least 1 h before the end of dialysis.
Time Frame: Baseline to 6 weeks
Population: The FAS population included all subjects who were randomised into the study, received at least one dose of the study drug, and had a Hb assessment. Subjects were included as randomised, regardless of which treatment they actually received.
Measure: Number; unit: percentage of participants
Arm/Group | Iron Isomaltoside 1000 | Iron Sucrose
Number analyzed (Participants) | 226 | 115
percentage of participants | 82.7 | 82.6

2. Secondary Outcome: Change in Hemoglobin Concentration
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: g/dL
Arm/Group | Iron Isomaltoside 1000 | Iron Sucrose
Number analyzed (Participants) | 216 | 113
g/dL | -0.07 [-5.5 to 2.9] | -0.06 [-4.9 to 2.8]

ADVERSE EVENTS:
Description: The safety population included all subjects who were randomised and received at least one dose of iron isomaltoside 1000 or iron sulphate. The safety analyses was performed on the safety population
Arm/Group | Iron Isomaltoside 1000 | Iron Sucrose
Serious Adverse Events (participants affected / at risk) | 22/230 | 6/114
Other Adverse Events (participants affected / at risk) | 42/230 | 16/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iron Isomaltoside 1000 (N=230) | Iron Sucrose (N=114)
acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
gingivalbleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
puncture site haemorrhage (General disorders) | 1 (1) | 0 (0)
sudden death (General disorders) | 1 (1) | 0 (0)
biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
arteriovenous fistula site infection (Infections and infestations) | 1 (1) | 0 (0)
device related infection (Infections and infestations) | 1 (1) | 0 (0)
infected fistula (Infections and infestations) | 1 (1) | 0 (0)
lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
staphylococcol bacteraimia (Infections and infestations) | 0 (0) | 1 (1)
fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
anaesthetic complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
brain stem infarction (Nervous system disorders) | 1 (1) | 0 (0)
nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iron Isomaltoside 1000 (N=230) | Iron Sucrose (N=114)
diarrhoea (Gastrointestinal disorders) | 5 (5) | 2 (2)
nasopharyngitis (Infections and infestations) | 6 (6) | 1 (1)
lower respiratory tract infection (Infections and infestations) | 4 (5) | 3 (4)
fall (Injury, poisoning and procedural complications) | 7 (7) | 0 (0)
procedural hypotension (Injury, poisoning and procedural complications) | 5 (18) | 1 (2)
C-reactive protein increased (Investigations) | 6 (6) | 1 (1)
hyperphosphataemia (Metabolism and nutrition disorders) | 5 (5) | 4 (4)
pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6) | 0 (0)
headache (Nervous system disorders) | 7 (7) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If Pharmacosmos or its agents has not prepared a draft for submission to a peer reviewed journal prior to 1 year following completion of the study report, the investigators have the right to publish the results. Such publications are to be submitted to Pharmacosmos for comment 30 days prior to submission for publication.